CLINICAL TRIAL: NCT00349115
Title: Induction Therapy With TCD Regimen (Thalidomide, Cyclophosphamide, Dexamethasone) Followed by Autologous Stem Cell Transplantation in Newly Diagnosed Multiple Myeloma Patients
Brief Title: TCD Followed by autoSCT for Newly Diagnosed MM Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Multiple Myeloma Working Party (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Korean Multiple Myeloma Working Party
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMM53
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2006-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
Multiple Myeloma is a incurable disease. Thalidomide in combination with other agents are currently in trials for the newly diagnosed patients, we designed treatment of TCD, followed by high dose chemotherapy with autologous stem cell transplantation and TD maintenance therapy for the patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
Phase II clinical trial for the patients with newly diagnosed. TCD (thalidomide, cyclophosphamide and dexamethasone) will be applied for the patients as an induction chemotherapy, followed by high dose chemotherpy and autologous stem cell transplantation. Afterthen, they will receive TD (thalidomide and dexamethasone) maintenance therapy for one year.

ELIGIBILITY:
Inclusion Criteria:Newly diagnosed multiple myeloma in aged between 18 and 75 years old with following mesurable leisons: (serum M-protein ≥ 1 g/dL or urine M-protein ≥ 400 mg/day) -

Exclusion Criteria:

- 1. Smoldering or indolent myeloma 2. ECOG performance status > 3 point 3. Known hypersensitivity to cyclphosphamide, thalidomide or dexamethasone 4. Peripheral neuropathy or neuropathic pain Grade 2 or higher as defined by NCI CTCAE version 3 5. Uncontrolled or severe cardiovascular disease, including MI within 6 months of enrolment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis, cardiac ejection fraction <0.5 : Severe conduction disorder : Hypotension (sitting systolic BP ≤ 100 mmHg and/or sitting diastolic BP ≤ 60 mmHg 6. Impaired hepatic function (AST or ALT ≥ x 3 upper normal, T-bilirubin ≥ x 2 upper normal) 7. Creatinine cliearance < 20 ml/min 8. Corrected serum calcium ≥ 14 mg/dL 9. Sepsis or current active infection 10. Pregnancy or breast feeding 11. Uncontrolled Diabetes Mellitus 12. Previous history of Recurrent DVT or pulmonary embolism 13. Active ulcers detected by gastroscopy 14. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

15. Receipt of extensive radiation therapy within 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2006-06; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Response rate of TCD induction Therapy

SECONDARY OUTCOMES:
Progression free survival and Overall survival of TCD, followed by high dose chemotherapy and autoPBSCT and TD maintenance
To evaluate toxicities of TCD, followed by high dose chemotherapy and autoPBSCT and TD maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Je-Jung Lee, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Je-Jung Lee, Hwsun-eup, Hwasun-gun, Jeollanam-do, South Korea